CLINICAL TRIAL: NCT01508286
Title: Multicenter, Open-label, Early Access Program of Telaprevir in Combination With Peginterferon Alfa and Ribavirin in Genotype 1 Chronic Hepatitis C Subjects With Severe Fibrosis and Compensated Cirrhosis
Brief Title: Early Access Program of Telaprevir With Peginterferon and Ribavirin in Chronic Hepatitis C Subjects
Status: No longer available | Type: Expanded Access
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017857; VX-950HEP3002 (Other: Janssen); 2010-023669-23 (EudraCT Number)
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C
Keywords: telaprevir; hepatitis C; early access program
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin

INTERVENTIONS:
Drug: Telaprevir + peginterferon alfa + ribavirin — During the first 12 weeks of the early access program, all eligible patients will receive telaprevir 750 mg every 8 hours in combination with peginterferon-alfa and ribavirin.
  Other Names: experimental
Drug: peginterferon alfa + ribavirin — Patients with severe fibrosis who are treatment naïve or prior treatment relapsers will subsequently be treated with peginterferon-alfa and ribavirin alone for either an additional 12 or 36 weeks.
  Other Names: experimental
Drug: peginterferon alfa + ribavirin — Previously treated patients with prior partial or null response, or who had viral breakthrough, with severe fibrosis and all subjects with cirrhosis will subsequently be treated with peginterferon-alfa and ribavirin alone for an additional 36 weeks.
  Other Names: experimental

SUMMARY:
The purpose of this early access program is to provide telaprevir to patients with a specific type of hepatitis C viral infection (termed 'genotype 1') who are expected to benefit from telaprevir-based therapy but who reside in countries in which telaprevir is not yet commercially available and who are not eligible for enrollment into a clinical study of telaprevir. The study also aims to collect information on the safety and adverse events with telaprevir treatment in combination with peginterferon alfa and ribavirin, which is typically used to treat patients with hepatitis C. In addition to hepatitis C viral infection, patients in this study will also have a diagnosis of liver fibrosis and compensated liver disease.

DETAILED DESCRIPTION:
This is a multicenter, multinational, open-label, non-comparative early access program designed to provide telaprevir to patients infected with hepatitis C virus genotype 1, who have a documented diagnosis of liver fibrosis and compensated liver disease (Child Pugh Grade A), and are expected to benefit from telaprevir-based therapy. Patients will be excluded if they are eligible for enrollment into an ongoing clinical study of telaprevir. Enrollment of patients into this study will continue until telaprevir becomes available for reimbursement in the country in which a patient resides or until September 2013, whichever occurs first, unless otherwise indicated per local regulations. During the first 12 weeks of the study, all patients will receive telaprevir administered orally with food every 8 hours in combination with peginterferon-alfa/ribavirin [PEG-IFN-alfa/RBV]). Patients will then be treated with Peg-IFN-alfa/RBV alone for an additional 12 or 36 weeks, based on how they respond to treatment (assessed by levels of hepatitis C viral RNA in the plasma, which reflects the number of virus particles in the bloodstream) and/or by type of patient (patients with severe fibrosis who had not received prior treatment or had previously relapsed during treatment, patients with prior partial or null response [who had only partially or had not responded to previous treatment], patients who had viral breakthrough [recurrence of viral copies during antiviral treatment], or patients with cirrhosis). For all patients, rules will be applied to ensure that telaprevir or Peg-IFN-alfa/RBV are stopped if subjects have viral breakthrough or treatment failure. All patients should have a follow up visit (including measurement of hepatitis C viral RNA levels in the bloodstream) 24 weeks after the last administered dose of any treatment. Dose modifications of telaprevir are prohibited and once telaprevir treatment is discontinued it may not be reinitiated in this study.

ELIGIBILITY:
Inclusion Criteria:

* have evidence of hepatitis C virus infection genotype 1 (by molecular assay); - have quantifiable plasma hepatitis C viral RNA levels; - have documented liver fibrosis as assessed by liver biopsy or a non-invasive test showing severe fibrosis or cirrhosis (for subjects with severe fibrosis, the diagnostic test should have been performed within the past 18 months); - have compensated liver disease (Child-Pugh Grade A clinical classification); - have access to hepatitis C treatment (peginterferon-alfa/ribavarin)

Exclusion Criteria:

* eligible for enrollment into an ongoing clinical study of telaprevir; - infected or co-infected with hepatitis C virus of a genotype other than genotype 1 and/or co-infected with HIV; - contraindication to the administration of peginterferon-alfa or ribavarin, or medical history or laboratory values that preclude treatment with peginterferon-alfa or ribavarin according to the respective local prescribing information; - history of having previously received an investigational treatment with hepatitis C viral protease or polymerase inhibitors (a class of drugs like telaprevir); - signs or symptoms of hepatocellular carcinoma (tests for serum alpha-fetoprotein and ultrasonography should have been done a maximum of 4 months before screening to screen for hepetocellular carcinoma)

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (128):
- Australia (22):
  - Adelaide
  - Bedford
  - Box Hill
  - Camperdown
  - Central Queensland M C
  - Concord
  - Darlinghurst
  - Fitzroy
  - Fremantle
  - Greenslopes
  - Heidelberg
  - Herston
  - Kingswood
  - Kogarah
  - Liverpool
  - Melbourne
  - New Lambton Heights
  - Parkville
  - Parkville - Vic
  - Perth
  - Sydney
  - Woolloongabba
- Austria (5):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
  - Wels
- Belgium (9):
  - Antwerp
  - Bruges
  - Brussels
  - Edegem
  - Genk
  - Ghent
  - Laken (Brussel)
  - Leuven
  - Liège
- Brazil (5):
  - Pinheiros
  - Porto Alegre
  - Recife
  - Rio de Janeiro
  - São Paulo
- Czechia (5):
  - Hradec Králové
  - Opava
  - Prague
  - Praha 4 N/A
  - Ústí nad Labem
- Germany (13):
  - Berlin
  - Cologne
  - Düsseldorf
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - Herne
  - Leipzig
  - München
  - Münster
  - Würzburg
- Greece (8):
  - Alexandroupoli
  - Athens
  - Heraklion Crete
  - Ioannina
  - Larissa
  - Pátrai
  - Thessaloniki
  - Thessalonikis
- Hungary (7):
  - Budapest
  - Debrecen
  - Gyula
  - Kaposvár
  - Pécs
  - Szeged
  - Székesfehérvár
- Luxembourg, Luxembourg
- New Zealand (3):
  - Auckland
  - Christchurch
  - Hamilton
- Romania (5):
  - Bucharest
  - Constanța
  - Iași
  - Ploieşti
  - Timișoara
- Russia (6):
  - Moscow
  - Saint Petersburg
  - Samara
  - Stavropol
  - Tyumen
  - Yekaterinburg
- Serbia (4):
  - Belgrade
  - Belgrade Serbia
  - Niš
  - Novi Sad
- Spain (27):
  - A Coruña
  - Alcorcón
  - Alicante
  - Almería
  - Ávila
  - Barakaldo
  - Barcelona
  - Córdoba
  - Donostia / San Sebastian
  - Girona
  - Granada
  - La Coruÿa N/A
  - León
  - Madrid
  - Majadahonda (Madrid)
  - Málaga
  - Oviedo
  - Palma de Mallorca
  - Pamplona
  - Pontevedra
  - Sabadell
  - Santa Cruz de Tenerife
  - Santander
  - Seville
  - Toledo
  - Valencia
  - Zaragoza
- Switzerland (8):
  - Basel
  - Basel Bs
  - Bern
  - Geneva
  - Lausanne
  - Lugano
  - Sankt Gallen
  - Zurich

REFERENCES:
- [Derived] Lepida A, Colombo M, Fernandez I, Abdurakhmanov D, Ferreira PA, Strasser SI, Urbanek P, Mangia A, Calleja JL, Iraqi W, DeMasi R, Lonjon-Domanec I, Moreno C, Wedemeyer H. Final Results of the Telaprevir Access Program: FibroScan Values Predict Safety and Efficacy in Hepatitis C Patients with Advanced Fibrosis or Cirrhosis. PLoS One. 2015 Sep 23;10(9):e0138503. doi: 10.1371/journal.pone.0138503. eCollection 2015. PMID 26398503
- See also: Multicenter, Open-Label, Early Access Program of Telaprevir in Combination With Peginterferon Alfa and Ribavirin in Genotype 1 Chronic Hepatitis C Subjects With Severe Fibrosis and Compensated Cirrhosis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2490&filename=CR017857_CSR.pdf